CLINICAL TRIAL: NCT06275815
Title: Promoting Caregiver Implementation of an Effective Early Learning Intervention: Sit Together and Read (STAR)
Brief Title: Promoting Caregiver Implementation of an Effective Early Learning Intervention
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: Nationwide Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: R01DC020958 (NIH)
Record Dates: First submitted 2024-01-29; First posted 2024-02-23 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Developmental Language Disorder; Reading; Difficult
Keywords: Randomized Control Trial; Print Knowledge; Reading Outcomes; literacy; behavior-change strategies; early literacy
MeSH Terms: conditions — Language Development Disorders; Dyslexia; Literacy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Untreated Control (No Intervention): Caregivers read to child as usual over 15 week period.
- STAR Only (Experimental): Typical implementation of Sit Together and Read (STAR)
  Interventions: Other: Sit Together and Read (STAR)
- STAR + Reward (Experimental): Typical implementation of Sit Together and Read (STAR) plus additional small monetary incentives for caregivers
  Interventions: Other: Sit Together and Read (STAR); Behavioral: Monetary Reward
- STAR + text encouragement (Experimental): Typical implementation of Sit Together and Read (STAR) plus caregivers receive encouraging text messages
  Interventions: Other: Sit Together and Read (STAR); Behavioral: Text Encouragement

INTERVENTIONS:
Other: Sit Together and Read (STAR) — Sit Together and Read (STAR) features an explicit, systematic sequence of 15 objectives that target four dimensions of print knowledge: print organization, print meaning, letters, and words. These objectives are explicitly targeted in the context of repeated adult-child shared reading sessions and are systematically cycled over an intervention period so the child has repeated opportunities for acquiring the targeted print objectives. STAR is a manualized 15-week intervention.
  Other Names: STAR Read-Aloud Practices; Read-Aloud Practices
  Arms: STAR + Reward; STAR + text encouragement; STAR Only
Behavioral: Monetary Reward — Caregiver receives a monetary reward of $0.50 for each session logged (up to 60 sessions) and audio-recording completed (up to 15 audio recordings).
  Arms: STAR + Reward
Behavioral: Text Encouragement — Caregiver receives three tailored encouraging text messages specific to each week of the Sit Together and Read intervention.
  Other Names: SMS Messaging
  Arms: STAR + text encouragement

SUMMARY:
The goal of this study is to examine the impact of a caregiver-implemented shared reading program, Sit Together and Read (STAR), on children ages 4 to 5 with developmental language disorder. The main questions it aims to answer are:

* how much STAR impacts children's literacy skills in the short-term and long-term--up to two-years after completing STAR.
* how do caregiver supports in the form of small monetary rewards or encouraging texts help caregivers to implement STAR at its intended frequency of sessions per week.

Caregiver participants will be assigned to either a control group or one of three STAR groups. Children's skills related to literacy and learning will be assessed before the intervention starts, at the end of the intervention, and every six months post-intervention for two years.

Researchers will determine the short term and long term impacts of STAR compared to the control group. Researchers will compare the three STAR conditions to see if the rewards or encouragement helped parents to follow through with completing more STAR sessions.

ELIGIBILITY:
Inclusion Criteria:

* receiving or on waitlist for speech services
* primary complaint of impaired language skills
* receptive, expressive, or mixed language disorder
* primarily communicates in English

Exclusion Criteria:

1. No known additional diagnoses causal of developmental language disorder including

   1. autism spectrum disorder
   2. hearing loss
   3. severe intellectual disability
2. Is not attending or has completed Kindergarten

Ages: 48 Months to 71 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 320 (Estimated)
Dates: Start 2024-04-10 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Preschool Word and Print Awareness (PWPA) | Pretest before intervention and post-test immediately following intervention
  Standardized criterion-referenced measure of children's knowledge of 15 basic print concepts
Phonological Awareness Literacy Screening (PALS): Alphabet Knowledge and Name Writing | Pretest before intervention and post-test immediately following intervention
  PALS-Preschool is a scientifically-based phonological awareness and literacy screening and progress measure that assesses preschoolers' developing knowledge of important literacy fundamentals. The assessment reflects skills that are predictive of future reading success. We administer two subtests that measures name writing ability and upper-case and lower-case alphabet recognition.
The Reading House (THR) | Pretest before intervention and post-test immediately following intervention
  A direct screening tool developed for use with pediatricians that allows a variety of providers to identify children who may be at risk for reading difficulties. It is a direct, book-based screener grounded in the concept of emergent literacy. TRH assessment examines 1) print knowledge, 2) alphabet knowledge, 3) letter-sound knowledge, 4) phonological awareness, 5) vocabulary, and 6) emergent writing.
Woodcock Johnson Test of Achievement- IV (WJ-IV): Word Attack and Letter-Word Identification | Completed at all assessing timepoints. Pretest, immediate post-test, 6 month follow-up, 12 month follow-up, 18 month follow-up, 24 month follow up.
  We administer two subtests of the norm referenced, standardized WJ-IV, Word Attack and Letter-Word Identification. Measure of child literacy and reading skill. We will explore avenues for data reduction, including use of a latent-variable modeling strategy.
Woodcock Johnson Test of Achievement- IV (WJ-IV): Spelling, Passage Comprehension | 6 month follow-up, 12 month follow-up, 18 month follow-up, 24 month follow up.
  We administer two subtests of the norm referenced, standardized WJ-IV, Spelling and Passage Comprehension. Measure of child literacy and reading skill

CONTACTS AND LOCATIONS:
Overall Officials: Laura M Justice, PhD, Principal Investigator — Ohio State University
Locations (2):
- United States (2):
  - Schoenbaum Family Center; Crane Center for Early Childhood Research and Policy, Columbus, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio